CLINICAL TRIAL: NCT06401798
Title: Radiographic and Clinical Assessment of Locally Delivered Camel Whey Protein Gel and Camel Whey Protein Nanoparticles Gel in Stage II Grade B Periodontitis: Randomized Controlled Clinical Trial.
Brief Title: Locally Delivered Whey Protein Nanoparticles Gel in Stage II Grade B Periodontitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Walid Elamrousy, Assistant Professor of periodontology, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KFSIRB200-189
Record Dates: First submitted 2024-05-02; First posted 2024-05-07 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Periodontitis Chronic Localized Slight

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- placebo control group (Placebo Comparator): After proper scaling and root planning, placebo gel will be applied topically to the affected sites.
  Interventions: Drug: placebo gel
- CWP group (Active Comparator): Topical application of CWP gel will be applied topically to the affected sites.
  Interventions: Drug: CWP gel
- NCWP group (Active Comparator): CWP nanoparticles gel will be applied topically to the affected sites.
  Interventions: Drug: NCWP gel

INTERVENTIONS:
Drug: placebo gel — Methylcellulose gel was applied topically to the pocket
  Other Names: Methylcellulose gel
  Arms: placebo control group
Drug: CWP gel — Methylcellulose gel combined with CWP was applied topically to the pocket
  Other Names: Camel Whey Protein
  Arms: CWP group
Drug: NCWP gel — Methylcellulose gel combined with NCWP was applied topically to the pocket
  Other Names: Nano-Camel Whey Protein
  Arms: NCWP group

SUMMARY:
Aim of the current study is to evaluate radiographic and clinical alterations following topical application of CWP gel and CWP nanoparticles gel in stage II grade B periodontitis patients.

DETAILED DESCRIPTION:
Periodontal disease is an oral inflammatory process that is typically initiated by bacterial infection stimulating the host response to produce various inflammatory mediators in high levels, which are also involved in the initiation and progression of periodontal disease.Such mediators generate a cascade reaction that eventually leads to the irreversible degradation of connective tissues and bone, with subsequent loss of periodontal attachment.

A new periodontitis classification scheme has been adopted, in which forms of the disease previously recognized as "chronic" or "aggressive" are now grouped under a single category ("periodontitis") and are further characterized based on a multi-dimensional staging and grading system. Staging is largely dependent upon the severity of disease at presentation as well as on the complexity of disease management, while grading provides supplemental information about biological features of the disease including a history-based analysis of the rate of periodontitis progression; assessment of the risk for further progression; analysis of possible poor outcomes of treatment; and assessment of the risk that the disease or its treatment may negatively affect the general health of the patient. periodontitis is classified using a system of staging and grading:

Staging reflects the severity and extent of disease based on tissue destruction:

* Stage I: Interdental CAL 1-2 mm, no tooth loss due to periodontitis, maximum probing depth ≤4 mm with horizontal bone loss mostly.
* Stage II: Interdental CAL 3-4mm, no tooth loss due to periodontitis, maximum probing depth ≤5mm with horizontal bone loss mostly.
* Stage III: Interdental CAL ≥5 mm, tooth loss due to periodontitis of ≤4 dents, maximum probing depth ≥ 6 mm and mostly associated with vertical bone loss.
* Stage IV: Interdental CAL ≥5 mm, tooth loss due to periodontitis of ≥5 dents and maximum probing depth ≥ 6 mm.

Grading of periodontitis refers to how quickly the disease is progressing.

* Grade A (Slow): Bone loss is progressing slowly.
* Grade B (Moderate): Bone loss is progressing at a moderate rate.
* Grade C (Rapid): Bone loss is progressing rapidly. The ultimate goal of periodontal therapy is to prevent further disease progression in order to reduce the risk of tooth loss and to restore the tissues that have been lost as a result of periodontitis. (4) The gold-standard treatment for periodontitis is subgingival debridement associated with effective supragingival biofilm control. However, even though mechanical debridement presents favorable short-term results, these benefits may not be maintained in the long-term, especially in susceptible individuals who develop a chronic (hyper)inflammatory response against the microbiome that is associated with genetic, systemic, or environmental factors. Failure of periodontal therapy stems largely from an inability to re-verse biofilm dysbiosis and to control inflammation. Therefore, antimicrobial agents and immune modulators have been considered for the treatment of periodontitis.

The additional use of antibiotics, systemically in the treatment of periodontitis is limited, due to the need for high doses to achieve the appropriate concentration of the drug in the gingival fluid, rapidly growing resistance of the bacteria, and side effects of the drugs. In addition, due to the advanced organization of the structure and function of the subgingival biofilm, antibiotics may not be effective or can be inactivated. Therefore, for almost 30 years, drug systems (antibiotics, antiseptics anti-inflamatories and anti-oxidants) have been developed in the form of direct subgingival administration. The advantage of this form of treatment is the significant concentration of the drug after application and its persistence for up to several weeks. With this form of application, many side effects that are associated with general systemic therapy can be avoided.

Camel whey protein (CWP) has a potent natural antioxidative effect as it reduces the oxidative stress and strengthens the immune system functions. The beneficial effects of CWP dietary supplementation include the stimulation of adaptive and innate immunity and anti-inflammatory, antibacterial, anticancer, antiviral, and antioxidative effects In addition, it has been shown that CWP improves the treatment of impaired wound healing in diabetic patients. Studies have demonstrated the consequences of supplementary CWP on the reduction of inflammatory biomarkers, proinflammatory cytokines, modulation of the immune functions, and free radicals' reactive oxygen species. Those effects of CWP could play a potential role in treating periodontitis.

Local delivery of nanoparticles emerges as a promising strategy for improved treatment. These nanoparticles, due to their minute size and tailorable properties, offer targeted drug delivery to the periodontal pocket. This approach concentrates therapeutic effects at the infection site, potentially enhancing treatment efficacy while minimizing systemic side effects of conventional medications.

Due to technical developments and the availability of cone-beam computed tomography (CBCT), 3-D imaging has become feasible and offers some advantages and potential for the evaluation of complex anatomical structures. CBCT illustrates and validates the possibility of radiographically visualizing and metrically assessing hard and soft periodontal tissues.

No previous researches have examined the outcomes of CWP on the treatment of periodontitis. Consequently, the current study was designed to assess the effects of topical CWP gel and CWP nanoparticle gel as an adjunct to nonsurgical therapy versus nonsurgical therapy alone on the clinical as well as radiographic parameters of stage II grade B periodontitis patients.

ELIGIBILITY:
Inclusion Criteria:

* patients will be selected to be systemically free with stage II periodontitis
* having 3-4 mm interdental clinical attachment loss (CAL) at ≥2 nonadjacent teeth
* maximum probing depth ≤5 mm

Exclusion Criteria:

* smokers
* pregnant and lactating females
* patients received any type of periodontal treatment in the past 6 months prior to examination
* patients who used antibiotic or anti-inflammatory drugs or antioxidants within the 6 months preceding the beginning of the study

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2024-05-05 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-03-15 (Actual)

PRIMARY OUTCOMES:
Bone height: | 6-months
  This incorporated the measurement of the bone defect height from the cemento-enamel junction (CEJ) to the base of the defect BD, the level of the alveolar crest from CEJ to the alveolar crest (AC), the bone defect depth from AC to BD). A line perpendicular was drawn from the AC to the root surface, and the intersection point across the root surface was considered as AC. The distance from the point AC to the base of the defect (AC-BD) will be considered as the intraosseous defect depth.
Mesiodistal (MD) and buccolingual (BL) bone defect width | 6-months
  The distance from the point AC to the alveolar crest (AC) will be considered as the MD width of the intraosseous defect. The BL width will be measured in the axial plane as the horizontal distance between the most coronal point for the buccal and lingual alveolar crest. A slice thickness of 0.2 mm will be used for CBCT analysis

CONTACTS AND LOCATIONS:
Overall Officials: Walid AH ELAMROUSY, PhD, Principal Investigator — Kafrelsheikh University
Locations (1):
- oral medicine and periodontology outpatient clinic, faculty of dentistry, kafrelsheikh University, Kafr ash Shaykh, Kafrelsheikh, Egypt

IPD SHARING:
Plan to Share IPD: No